CLINICAL TRIAL: NCT05725564
Title: PCORI-HA-2021C3-25041 Comparative Effectiveness of Brief Strength and Balance Exercises and Standard Home-Based Group Exercise for Primary Care Patients With Mobility Disability
Brief Title: Testing Interventions for Mobility Through Exercise (TIME)
Acronym: TIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HA-2021C3-25041; PCORI-HA-2021C3-25041 (Other: PCORI)
Record Dates: First submitted 2023-01-12; First posted 2023-02-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Walking, Difficulty; Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FAST-BCT (Experimental): FAST exercise intervention without behavior change techniques applied. Daily exercise intervention including functional resistance training and personalized coaching.
  Interventions: Behavioral: FAST (Functional Activity Strength Training)
- FAST+BCT (Experimental): FAST exercise intervention with behavior change techniques applied. Daily exercise intervention including functional resistance training and personalized coaching with added reminders, education, goal setting, self monitoring, and feedback to encourage adherence and effort.
  Interventions: Behavioral: FAST (Functional Activity Strength Training); Behavioral: Behavioral Change Technique
- BT-BCT (Active Comparator): Band Together exercise intervention without behavior change techniques applied. 3 times weekly group exercise intervention held over Zoom featuring strength and balance exercises for 45 minutes.
  Interventions: Behavioral: Band Together
- BT+BCT (Active Comparator): Band Together exercise intervention with behavior change techniques applied. 3 times weekly group exercise intervention held over Zoom featuring strength and balance exercises for 45 minutes with added reminders, education, goal setting, self monitoring, and feedback to encourage adherence and effort.
  Interventions: Behavioral: Band Together; Behavioral: Behavioral Change Technique

INTERVENTIONS:
Behavioral: FAST (Functional Activity Strength Training) — Daily exercise intervention including functional resistance exercises and personalized coaching.
  Arms: FAST+BCT; FAST-BCT
Behavioral: Band Together — 3 times weekly group exercise over Zoom featuring strength and balance exercises for 45 minutes
  Arms: BT+BCT; BT-BCT
Behavioral: Behavioral Change Technique — Reminders, education, goal-setting, self-monitoring, and feedback used to encourage participants to increase effort and adherence
  Arms: BT+BCT; FAST+BCT

SUMMARY:
In this project, the team plans to test the impact of FAST, its brief home-based strength training program which includes performance goal setting, to a program for home (BAND TOGETHER) that is similar to one offered by Silver Sneakers, available online to millions of older adults, and includes strength, balance, and aerobic exercises. The team hypothesizes that the brief program (FAST) will improve leg function better than the standard program (BAND TOGETHER), by encouraging older adults to be more consistent with using it and to try harder when they do.

DETAILED DESCRIPTION:
One in four older adults, the fastest growing demographic group in the US, reports serious difficulty walking or climbing stairs. Older adults note that these walking difficulties "deprives you of your identity" and "affects my day to day life… I can't do very much work on my own." Walking difficulties impair people's quality of life more than depression, anxiety, or pain. Walking difficulties also increase the chances of future disability, death, and healthcare costs. Though strength training improves walking ability, fewer than one in five older adults do strength training enough to benefit. What is unknown is how to create a strength training program that improves the ability of older adults to walk and do other things they need and want to do and that older adults are willing to do.

One approach to designing a strength training program that has not been tried before is to make them shorter. In 2020, the project team set out to design a short strength training program that older adults could do at home that would improve their physical function and that they would consistently do. The program was called FAST (Functional Activity Strength Training) and, to make it more effective, the team set specific goals for how many additional repetitions each person should be able to do over 12 weeks. These goals were then mentioned repeatedly, and feedback was provided about how well people made progress toward these goals.

In the first study of FAST (FAST-1), 24 healthy older adults performed 30 seconds of squats and push-ups each day but received no personal supervision. Over six months, they performed the exercises on 73 percent of days, which led to large increases in the number of push-ups and squats they were able to do. In the second study of FAST (FAST-2), the team randomly assigned 97 older adults who had trouble walking, and those assigned to do 30 seconds each of chair stands and steps onto a stepper each day improved their ability to stand up from a chair and stand on one leg more than those who did not do the exercises.

In this project, the team plans to test the impact of FAST, its brief home-based strength training program which includes performance goal setting, to a program for home (BAND TOGETHER) that is similar to one offered by Silver Sneakers, available online to millions of older adults, and includes strength, balance, and aerobic exercises. The team hypothesizes that the brief program (FAST) will improve leg function better than the standard program (BAND TOGETHER), by encouraging older adults to be more consistent with using it and to try harder when they do.

This study will enroll 520 primary care patients who are at least 65 years of age and randomly assign them to have access to 12 months of daily FAST or three-times weekly BAND TOGETHER. Each program will be delivered via the internet and each patient will receive about 30 minutes per month of personal support. The study will enroll patients who have trouble walking, have access to the internet, can provide informed consent, and receive permission from their doctor. The study is designed to see whether patients who have access to FAST, after 12 months, have better walking ability, balance, and leg strength and can do their normal daily activities more easily and fall less often than patients who have access to BAND TOGETHER.

To help us understand how best to perform the study, as well as how best to share the results, the study team assembled a group of stakeholders that includes patients, primary care providers, fitness center directors, and people who work for insurance, public health, and senior services organizations. The team will bring those stakeholders together each year and consult them regularly to help make difficult decisions as they arise-decisions that may impact each group of stakeholders differently. Two patient partners will work with investigators to supervise the group of stakeholders and organize their feedback, structured as a public comment period, to help the research team make decisions that take into account the perspectives of all of the key groups of stakeholders involved in improving the physical function of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 65
* Self reported difficulty or inability to walk 1/4/ mile
* Access to the Internet
* Covid vaccination

Exclusion Criteria:

* Chest pain on the PAR-Q
* Participating in another research project involving physical activity, falls or weight loss
* Planning to move or have surgery in the next 12 months
* Cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 702 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Physical Function | 12 Months
  Patient-Reported Outcomes Measurement Scale (PROMIS-29). The minimum and maximum values are unable to do and without any difficulty, and a higher score means a better outcome.

SECONDARY OUTCOMES:
Lower Extremity Performance | 12 Months
  Short Physical Performance Battery. The minimum value is a score of 0 points, the maximum value is a score of 16. A higher score means a better outcome.
Dose Received | Through study completion, an average of 1 year
  Sessions completed per week (percent)
Effort (Rating of Perceived Exertion) | Monthly up to 12 months
  Rating of Perceived Exertion. The minimum value is 0 (at rest) and the maximum value is 10 (maximal). This is a purely subjective measure here a higher or lower score doesn't necessarily lead to a better outcome, but for our exercise study we have a target RPE of 5 for exercise.
Gait Speed (10 meter walk test) | 12 Months
  Gait Speed (10 meter walk test). Participants undergo two trials (comfortable speed and fast speed), and an average of the two trials is used as the gait speed in m/s.
Muscle Strength | 12 Months
  Upper and lower extremity strength
Walking Ability | 12 Months
  6 Minute Walk Distance
Fatigue, Pain | 12 Months
  Patient Reported Outcomes Measurement Scale (PROMIS-29). The minimum value for the fatigue scales is "not at all", the maximum value is "very much". A lower score means a better outcome. The minimum values for the pain scales are "not at all" and 0, the maximum values "very much" and 10. A lower value means a better outcome.
Falls | 12 Months
  Percent experiencing a fall-related injury
Physical Activity | 12 months
  Accelerometry over 7 days
Number of participants with a self-reported injury due to physical activities | Monthly up to 12 months
  Injuries due to physical activities
Program Satisfaction | Monthly up to 12 months
  Net Promoter Score. The maximum value is 10 and the minimum value is 0. A higher value means a better outcome.

OTHER OUTCOMES:
Body Weight (kg) | 12 Months
  Body Weight (kg)
Height (cm) | 12 Months
  Height (cm)
Sociodemographics, self-reported medical history and tobacco use | Baseline
  Age, gender, race and ethnicity, medical history, smoking status, and education
Caregiving Status Questions (Receiving and Providing) | Monthly up to 12 months
  Giving and receiving caregiving, paid or unpaid, for personal care needs, such as eating, bathing, dressing, or getting around inside the home.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States